CLINICAL TRIAL: NCT02533323
Title: Phase 2 Trial of Pegaspargase-Gemox Chemotherapy in Newly Diagnosed, Nasal Type, Extranodal Natural Killer/T-cell Lymphoma
Brief Title: P-Gemox Regimen as First-line Chemotherapy in NK/T Lymphoma Patiens
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, dr. luyue, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-NK/T-5010
Record Dates: First submitted 2015-08-24; First posted 2015-08-26 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2016-10

CONDITIONS: Lymphoma, Extranodal NK-T-Cell
Keywords: NK/T-cell lymphoma; induction chemotherapy; survival
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Gemcitabine; Oxaliplatin; pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- P-Gemox (Experimental): P-Gemox:gemcitabine :1250mg/m2 (ivdrip) on days 1, oxaliplatin :85 mg/m2 (ivdrip) on day 1, and pegaspargase : 2500 IU/m2 (intramuscular injection) on day 1.Cycle is repeated every 14 days.
  Interventions: Drug: gemcitabine; Drug: oxaliplatin; Drug: pegaspargase

INTERVENTIONS:
Drug: gemcitabine — gemcitabine :1250mg/m2 (ivdrip) on days 1
  Other Names: Gemzar
Drug: oxaliplatin — oxaliplatin :85 mg/m2 (ivdrip) on day 1
  Other Names: Eloxatin
Drug: pegaspargase — pegaspargase : 2500 IU/m2 (intramuscular injection)
  Other Names: Oncaspar

SUMMARY:
This prospective study was conducted to evaluate the efficacy and safety profiles of first-line combined gemcitabine, oxaliplatin, and Pegaspargase (P-Gemox) in newly diagnosed, nasal type, extranodal natural killer/T-cell lymphoma.

DETAILED DESCRIPTION:
Treatment P-Gemox dosages were as follows: days 1, 30 min intravenous infusion of 1250 mg/m2 gemcitabine; day 1, 2h intravenous infusion of 85 mg/m2 oxaliplatin; day 1, deep intramuscular injection of 2500 U/m2 PEG-ASP at three different sites. The regimen was repeated every 2 weeks for a maximum of six cycles. Stage IE/IIE patients underwent four cycles induction chemotherapy, followed by involved-field radiotherapy after got CR, PR or SD. Three-dimensional conformal radiotherapy was done by linear accelerator at 2.0 grays (Gy) per daily fraction with 5-6 weeks. The involved- field radiation (IFRT) dose was 50-56 Gy. Stage IIIE/IVE patients patients underwent at least two cycles treatments unless there was disease progression or unacceptable side effects, or withdrawal of patient consent. Primary tumor radiotherapy was recommended after they achieved CR.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed ENKTL
* age:18-80years
* at lease one measurable lesion
* receive no chemotherapy or radiotherapy before
* Eastern CooperativeOncology Group performance status of 0 to 2.
* Adequate hematologic function (eg, white blood cell ≥ 3×10e9/l,neutrophils count ≥1.5×10e9/L, and platelet count≥ 100×10e9/L),renal function (eg, serum creatinine≤1.5 mg/dL and creatinine clearance ≥50 mL minute), and hepatic function (e.g, total bilirubin≤ 2 times the upper limit of normal and aspartate and alanine transaminase levels ≤ 3 times the upper limit of normal)

Exclusion Criteria:

* mismatch the inclusion criteria
* systematic central nervous system involvement, previous or concomitant malignancies and any coexisting medical problems that could cause poor compliance with the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
progression free survival | up to end of follow-up-phase (approximately 3 years)
  time from the date of enrollment to date of disease progression, or death of any cause, or date of lost follow-up, whichever comes first

SECONDARY OUTCOMES:
complete remission rate | every 4 weeks,up to completion of treatment(approximately 6 months)
  The criteria for the efficacy evaluation (overall response rate and complete remission) of the regimen is according to the following article:
  Cheson BD, Horning SJ, Coiffier B, et al. Report of an international workshop to standardize response criteria for non-Hodgkin's lymphomas. NCI Sponsored International Working Group. J Clin Oncol. 1999;17:1244.
overall survival | up to end of follow-up-phase (approximately 3 years)
  overall survival (OS): time from the date of enrollment to date of death from any cause, or date of lost follow-up, whichever comes first
safety, as measured by adverse events | up to end of follow-up-phase (approximately 3 years)
  ncluding hematological safety and non-hematological safety.All the adverse events will be classified according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE)
serum soluble programmed death ligand 1 | every 3 weeks,up to completion of treatment(approximately 6 months)
  Soluble PD-L1 is measured using an enzyme-linked immunosorbent assay
serum interleukin 15 | every 3 weeks,up to completion of treatment(approximately 6 months)
  serum interleukin 15 is measured using an enzyme-linked immunosorbent assay
Serum ferritin level | every 3 weeks,up to completion of treatment(approximately 6 months)
  Serum ferritin level is measured using radioimmunoassay

CONTACTS AND LOCATIONS:
Overall Officials: yue lu, MD., Principal Investigator — Department of Hematological Oncology, Sun Yat-sen University Cancer Center
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China